CLINICAL TRIAL: NCT02338375
Title: Clinical Trial of the Safety and Efficacy of Allogenic Umbilical Cord Blood-derived Mesenchymal Stem Cell Product With Microfracture for Osteochondral Lesion of Talus Patients
Brief Title: Safety and Efficacy of Allogenic Umbilical Cord Blood-derived Mesenchymal Stem Cell Product
Acronym: Cartistem
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, ChulWon Ha, MD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-10-078
Record Dates: First submitted 2013-07-31; First posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Osteochondral Lesion of Talus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cartistem (Experimental): For control group patients currently standard treatment of arthroscopic curettage and microfracture is performed, and for study group patients allogenic umbilical cord blood-derived mesenchymal stem cell product(Cartistem®) is added on the lesion after above mentioned procedure.
  Interventions: Biological: Cartistem
- standard treatment (Active Comparator): standard treatment of arthroscopic curettage and microfracture for osteochondral lesion of talus
  Interventions: Biological: Cartistem

INTERVENTIONS:
Biological: Cartistem — Cartistem is allogenic umbilical cord blood-derived stem cell product. Cartistem is 500uL/cm2 applied according to the lesion.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of adding allogenic umbilical cord blood-derived stem cell product(Cartistem®) on currently standard treatment of arthroscopic curettage and microfracture for osteochondral lesion of talus.

DETAILED DESCRIPTION:
same as above

ELIGIBILITY:
Inclusion Criteria:

* Non-responder to conservative treatment for radiographically confirmed (by MRI) osteochondral lesion of talus with ankle pain and/or stiffness and less than 75 of the AOFAS score
* Age between 20 and 70 year-old
* Appropriate function of blood clot PT(INR) < 1.5, APTT <1.5×control
* Appropriate renal function Creatinine ≤ 2.0 ㎎/㎗, proteinuria less than trace with Dipstick urine test
* Appropriate hepatic function Bilirubin ≤ 2.0 ㎎/㎗, AST/ALT ≤ 100 IU/L
* No evidence of autoimmue disorder As screening test anti-nuclear antibody and/or anti-thyroglobulin antibody, if positive rheumatologist referral needed to confirm diagnosis
* No surgery or radiotherapy for the same ankle joint within 6 weeks
* Female patients agreeing with maintenance of contraception during study period
* No ligament instability greater than grade II (Grade 0 : none, Grade Ⅰ: 0~5㎜, GradeⅡ: 5~10㎜, Grade Ⅲ: >10㎜) with physical exam
* Patients agreeing with participation in this study and signed on informed consent by their own will

Exclusion Criteria:

* Degenerative ankle arthritis patients
* Patients with autoimmune disease
* Patients with infectious disease needed parenteral antibiotics
* Patients with myocardial infarction, congestive heart failure, other serious heart diseases or uncontrollable hypertion
* Patients with other serious medical illness
* Pregnancy or breast feeding patients
* Past history related with psychiatric illness or epilepsy
* Alcoholic abuse
* Heavy smoker
* Chronic inflammatory disease including rheumatoid arthritis
* Participants of other clinical trial within 4 weeks
* Patients treated with immunosuppressing agents such as Cyclosporin A or azathioprine within 6 weeks
* Unstable ankle joint(lesion site) greater than grade II at physical exam (Grade 0 : none, grade Ⅰ: 0~5㎜, GradeⅡ: 5~10㎜, Grade Ⅲ: >10㎜)
* Other inappropriate patients determined by the prinicipal investigator

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-12; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
evaluate the efficacy of adding allogenic umbilical cord blood-derived stem cell product(Cartistem®) by American Orthopaedic Foot and Ankle Society(AOFAS) HINDFOOT/ANKLE SCALE | Baseline, Week 4, Week 8, Week 12, Week 24, Week 48

SECONDARY OUTCOMES:
evaluate the efficacy of adding allogenic umbilical cord blood-derived stem cell product(Cartistem®) by 100-mm VAS(Visual Analogue Scale) | Baseline, Week 4, Week 8, Week 12, Week 24, Week 48

OTHER OUTCOMES:
evaluate the efficacy of adding allogenic umbilical cord blood-derived stem cell product(Cartistem®) by ICRS arthroscopic scale for repair of articular cartilage | Baseline, Week 4, Week 8, Week 12, Week 24, Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Gangnam-Gu, Seoul, South Korea